CLINICAL TRIAL: NCT01696890
Title: Integration of Follow-up by First and Second Line Practitioners Facilitated by Telemonitoring Versus Stand-alone Telemonitoring in Patients With Severe Heart Failure
Brief Title: Integration of Follow-up by First and Second Line Practitioners by Telemonitoring in Heart Failure.
Acronym: TEMA-HF2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of inclusions, sudden withdrawal of study coordinator
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Paul Dendale, Prof Dr, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEMAHF2
Record Dates: First submitted 2012-03-29; First posted 2012-10-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; telemonitoring; first line practitioners; integrated approach; efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- integrated care (Active Comparator): telemonitoring-assisted follow-up with intensive collaboration between general practitioner and specialized Heart failure clinic.
  Interventions: Device: integrated follow-up
- standard care (Active Comparator): telemonitoring- assisted follow-up with usual care by general practitioner, without supervision of heart failure clinic
  Interventions: Device: standard care

INTERVENTIONS:
Device: integrated follow-up — close interaction between HF clinic and general practitioner in response to telemonitoring alerts. All subjects will be monitored daily for heart rate, blood pressure, and body weight, after which these data are transferred automatically to the general practitioner. This device is custom-made.
  Arms: integrated care
Device: standard care — no interaction between HF clinic and general practitioner in response to telemonitoring alerts. General practitioner is responsible for adaptations to therapy according to clinical presentation of the patient.
  Arms: standard care

SUMMARY:
The aim of this study is to evaluate this model of telemonitoring-assisted close supervision and interaction between first and second line health professionals versus a model of telemonitoring without this integrated approach.

DETAILED DESCRIPTION:
The incidence of acute decompensated heart failure is increasing. Patients with severe heart failure are rehospitalised for decompensation several times each year, increasing the cost for health care. In these cases of recurrent decompensation, the medical intervention in hospital is often limited to increasing the dosage of diuretics or vasodilators until the patient reaches a compensated state. After discharge, a readmission can be expected within a few months. A multidisciplinary approach by primary physician, heart failure nurse, rehabilitation team and cardiologist has been shown to decrease rehospitalisation rate and increase quality of life.

Very recently, our study group showed that an intense collaboration between first line practitioner and heart failure clinic, facilitated by the use of telemonitoring, can reduce mortality and hospitalisation rate. This study was a RIZIV sponsored trial of 6 months follow-up in patients with chronic heart failure. However, a large randomised multicentre trial investigating the use of telemonitoring in a population of heart failure (NYHA II-III) patients did not find any difference between telemonitoring and usual care (Chaudry et al NEJM 2010). In contradiction with this study, a Cochrane meta-analysis (Ingliss 2010) in more than 5000 patients confirmed our finding with a reduction in mortality and morbidity. The question therefore remains which factors are responsible for success or failure of the use of telemonitoring. Based on our previous experience, the approach of close monitoring by telemonitoring, with first line intervention by the patient's general practitioner (GP) and supervision by the heart failure clinic, might be the critical success factor.

Therefore, the aim of this study is to evaluate this model of telemonitoring-assisted close supervision and interaction between first and second line health professionals versus a model of telemonitoring without this integrated approach.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for decompensation of systolic heart failure
* LVEF < 40% during hospitalization.

Exclusion Criteria:

* reversible forms of acute heart failure (acute ischemia, myocarditis,..)
* heart failure due to severe aortic stenosis
* participation in cardiac rehabilitation after discharge
* previous or actual residency in a nursing home
* creatinine clearance <15 ml/min
* planned dialysis in the next 6 months
* planned biventricular pacemaker or cardiac surgery
* life expectancy of less than 1 year due to other diseases
* severe obstructive pulmonary disease (Gold III)
* significant mental or cognitive problems interfering with the daily measurements or intake of medication.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
overall mortality | 6 months
number of rehospitalizations | 6 months
time investment by HF nurses | 6 months

SECONDARY OUTCOMES:
quality of life | 6 months
appearance of renal failure (glomerular filtration rate (GFR) <60 mL/min/1.73 m2) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: paul dendale, MD, PhD, Principal Investigator — Jessa Hospital
Locations (7):
- Belgium (7):
  - Middelheim Ziekenhuis, Antwerp
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria Middelares, Ghent
  - Jessa Hospital, Hasselt
  - AZ Groeninge, Kortrijk
  - Chr.Citadelle, Liège